CLINICAL TRIAL: NCT00647920
Title: Study of the Human Anti-TNF-Antibody Adalimumab
Brief Title: Study of Adalimumab Administered as Subcutaneous Injections in Adult Chinese Rheumatoid Arthritis Subjects Treated With Methotrexate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Michael Snyder/Clinical Research Manager, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M02-573
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 40 mg (Experimental)
  Interventions: Biological: adalimumab
- Placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: adalimumab — 40 mg adalimumab sc, every other week
  Other Names: ABT-D2E7; Humira
  Arms: 40 mg
Biological: placebo — placebo sc, every other week
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Study of the Adalimumab Administered as Subcutaneous Injections in Adult Chinese Rheumatoid Arthritis Subjects Treated with Methotrexate

ELIGIBILITY:
Inclusion Criteria:

* Meet ACR criteria for diagnosis of active RA and have at both screening and baseline visits 6 swollen joints and 9 tender joints.

Exclusion Criteria:

* A history of, or current, acute inflammatory joint disease of different origin than RA (e.g., mixed connective tissue disease, seronegative spondyloarthropathy, psoriatic arthritis, Reiter's syndrome, systemic lupus erythematosus or any arthritide with onset prior to age 16 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2003-07; Primary Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
ACR20 | Week 12

SECONDARY OUTCOMES:
ACR50 | Week 12
ACR70 | Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung, Taiwan

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778